CLINICAL TRIAL: NCT05559528
Title: Clinical Outcomes of Breast Cancer and Its Relation With Access to Health Care in Brazil: a Prospective Study in HER2-negative/Hormone Receptor-Positive Metastatic Disease
Brief Title: BRaziLian outcomE for metAStatic breasT Cancer
Acronym: BREAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital do Coracao (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: BREAST
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Breast Cancer; Breast Cancer Stage IV
Keywords: Breast Cancer; ER+/HER2-
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Public health system: Group with patients treated in the public health system in Brazil. They will be stratified according to whether or not CDK 4/6 inhibitors are used in therapy.
- Private health system: Group with patients treated in the private health system in Brazil. They will be stratified according to whether or not CDK 4/6 inhibitors are used in therapy.

SUMMARY:
Given the certain benefit in efficacy of adding CDK 4/6 inhibitor to first line endocrine therapy in metastatic breast cancer HR+ HER2- , the aim of this project is to evaluate whether patients without private health insurance may have worse outcomes than privately insured women due to limited access to such class of drugs during their treatments. Prospective observational study with 300 patients divided into two groups, one with patients from the public health system and the second with patients treated in the private service. Patients will be recruited in different regions of Brazil and will be followed for 24 months, stratified according to the use or not of the CDK 4/6 inhibitors.

DETAILED DESCRIPTION:
In Brazil, breast cancer is the most common carcinoma in women, non- melanoma skin carcinomas. 66,280 new cases of breast cancer were estimated for each year of the 2020-2022 triennium, which represents 29.7% of all cancers. It is the main cause of cancer death in women and mortality rates remain high due to the large number of cases diagnosed in advanced stages (around 40%).

According to data from Concord-3, five-year survival estimates in the country were 75.2% (73.9 - 76.5) for the period from 2010 to 2014. However, the 5-year survival rate in the same period was over 85% in 25 countries and reached approximately 90% in North America and Oceania (3). The survival rate in low- and middle-income countries is remarkably different.

This disparity in survival reflects the unequal access of the population to breast screening, difficulty in diagnosis, delayed treatment and limited access to first-line systemic therapy for advanced and metastatic tumors.

Notwithstanding, with the development of new, expensive drugs, breast cancer survival differences between Brazil and high-income countries may increase if the access to new agents is not assured.

One of the most important changes in the hormone positive breast cancer, recently identified, was the greatly increased function of proteins that stimulate cells to grow and multiply, known as CDK4 and 6 (Cyclin-Dependent Kinase). These are normal parts of the human cell, but in this type of tumor they work much faster than they should, making the tumor grow.

Recent studies showed benefit with new target therapies that lower recurrence and progression, as cyclin-dependent kinases 4 and 6 (CDK 4/6) inhibitors with endocrine therapies in hormone receptor (HR)-positive, human epidermal growth factor receptor 2 (HER2)- negative advanced breast cancer has shown substantial improvements in progression- free survival (PFS).

Palbociclib (IBRANCE®) is a first-in-class oral inhibitor of cyclin-dependent kinases 4 and 6 that blocks G1-to S-phase progression. There is a strong in-vitro and clinical evidence suggesting that the dual inhibition of CDK 4/6 and ER signaling is a highly effective therapeutic strategy in HR+ MBC. In the phase 2 PALOMA-1 trial, the addition of palbociclib to letrozole significantly improved progression-free survival in women with advanced estrogen receptor-positive and HER2-negative breast cancer. Subsequently, in the phase III trial that included postmenopausal patients with metastatic, HR-positive, HER2-negative breast cancer who had not received prior treatment for advanced disease, an improvement in PFS (24.8 vs. 14.5 months; hazard ratio [HR] 0.58, 95% CI 0.46-0.72) and objective response rate (ORR; 42 vs. 35 percent) was seen with the combination of palbociclib and letrozole compared with letrozole alone.

The National Comprehensive Cancer Network (NCCN) Panel recommends first line therapy for HR-positive HER2-negative with aromatase inhibitor (AI) in combination with CDK 4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) in postmenopausal women or premenopausal women receiving ovarian ablation or ovarian function suppression with an LHRH agonist, combinations of aromatase inhibitors with CDK 4/6 inhibitors (8). However, the situation is rather different in many countries, including Brazil, where the population has limited access to these medications.

The health system in Brazil is organized in two types of assistance: the public system, known as Unified Health System (SUS), where the policies and costs are regulated by the State, and a private system, where the coverage is regulated by the National Supplementary Health Agency (ANS) through agreements with health insurance plans. Nowadays, 75% of the Brazilian population is attended by the public system versus 25% in the Supplementary Health Service.

The commercialization of CDK 4/6 inhibitors was only released in the national territory in 2018, but until nowadays it is not accessible for the majority of patients. Of note, patients in the public health system do not gain access to this class of drugs and those with private insurances usually settle a lawsuit to obtain the treatment once CDK 4/6 inhibitors are not covered by the National Supplementary Health Agency.

Thus, the disparity in the access to these important treatments due to socioeconomic differences probably results in worse outcomes according to health care coverage.

ELIGIBILITY:
Inclusion Criteria:

* Women may be premenopausal or postmenopausal
* Metastatic advanced breast cancer
* ER-positive and/or PR-positive, HER2-negative tumor
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2 and 3.
* Start of first-line treatment from 2019

Exclusion Criteria:

* Localized or locally advanced disease
* Lack of information about hormonal receptor and HER2 status
* Breast cancer in men
* Breast cancer in pregnancy
* Have progressed from initiation of first-line treatment to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients with HR+ HER2 metastatic breast cancer divided into two groups: public health system and private service. Patients will be recruited from 20 cancer treatment centers (10 public and 10 private), chosen in different regions of Brazil. We estimate recruiting 20 patients from each private center and 40 patients from each public center, totaling 300 patients in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) is the time from the start of treatment to the date of event defined as the first documented progression or death due to any cause. According to RECIST criteria, progressive disease is defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.

SECONDARY OUTCOMES:
Overall Survival (OS) | 2 years
  Overall Survival (OS) is defined as the time from the date of first dose to the date of death due to any cause. Time Frame: Baseline up to approximately 36 months
Cost-effectiveness analysis (CEA) | 2 years
  Cost-effectiveness analysis (CEA) will be measured according to criteria of the World Health Organization. The direct medical costs used in the model will be the weighted average of the costs of the various procedures according to the perspective: a) SUS perspective: the DATASUS, SIGTAP, health price database and CMED price list will be considered e b) Supplementary Health Perspective - the ANS database and CMED price list will be considered
EQ-5D questionnaire | 2 years
  Quality of life will be evaluated by EQ-5D questionnaire is designed for self-completion and, as such, captures information directly from the respondent,however, in this research the questionnaire will be applied by telephone contact.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa M Sanvido, PhD, Principal Investigator — Hospital do Coracao; Afonso CP Nazário, Professor, Principal Investigator — Hospital do Coracao; Luciola B Pontes, MD, Principal Investigator — Hospital do Coracao
Locations (1):
- Hcor, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sanvido VM, Pontes LB, Machado RH, Gomes JO, Barbante LG, Nicola ML, Tokunaga SM, Miranda TA, Laranjeira LN, Negrelli KL, Valeis N, Moutinho MSP, Helber HA, Sa RDS, Kawano-Dourado L, Cavalcanti AB, Nazario ACP. Study protocol to assess clinical outcomes of breast cancer and its relationship with access to healthcare in Brazil-BREAST trial (BRaziLian outcomE for metAStatic breasT cancer): a prospective observational study in HER2-negative/hormone receptor-positive metastatic disease. BMJ Open. 2025 Jun 30;15(6):e087877. doi: 10.1136/bmjopen-2024-087877. PMID 40588378